CLINICAL TRIAL: NCT06245226
Title: Assessment of Posture, Balance, Gait Disorders in Patients With Fibromyalgia and Investigation of Their Relationships With Disease-related Parameters
Brief Title: Assessment of Posture, Balance, Gait Disorders in Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Baran Tuncer, Medical Doctor (Physical Medicine and Rehabilitation Resident Doctor), Ankara City Hospital Bilkent
Other Study IDs: 10025142
Record Dates: First submitted 2023-12-12; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Posture; Postural stability; Balance; Gait
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia group: 50 female fibromyalgia patients
- Control group: 50 pain-free female volunteers

SUMMARY:
The study aims to determine the posture, balance and gait disorders objectively in patients with fibromyalgia (FM) and to investigate their relationships with disease-related parameters.

DETAILED DESCRIPTION:
After being informed about study and potential risks, all participants giving written informed consent will undergo screening period determine eligibility for study entry. The participants who met the eligibility recruitments will get into the assessment.

The study will include 100 participants aged between 18-65 years and without any disease or orthopedic disorder that can cause posture, balance and gait disorders: 50 female patients who met the ACR (American College of Rheumatology) 2016 FM diagnostic criteria and 50 pain-free females.

Researcher will record sociodemographic data of all participants and disease duration of patients with FM. The researcher will evaluate disease activity by Fibromyalgia Impact Questionnaire, sleep quality by Pittsburgh Sleep Quality Index and fatigue severity by Fatigue Severity Scale in FM group.

In both groups the researcher will use; DIERS formetric 3D/4D video-rasterstereography (Diers International GmbH, Schlangenbad, Germany) device for the posture analyze, HUR SmartBalance BTG4 system (Hur Labs, Kokkola, Finland) for postural balance control and limits of stability measurements, Zebris FDM type 3 (Zebris Medical GmbH, Germany) gait analysis system for measuring spatio-temporal gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Fibromyalgia according to ACR 2016 diagnostic criteria
* Signing written informed consent to participate in the study

Exclusion Criteria:

* Rheumatological, neurological and/or psychiatric diseases that may cause balance and gait disorders (cerebrovascular accident sequelae, Parkinson's, myasthenia gravis, polyneuropathy, rheumatoid arthritis, ankylosing spondylitis, major depression)
* Other diseases that cause balance and other gait disorders (history of major trauma to the lower extremity, and/or orthosis users, those who have had spinal and/or lower extremity surgery)
* Orthopedic disorders that may cause limitation in joint range of motion and/or loss of motor muscle strength
* Those who cannot take commands due to cognitive dysfunction
* Vestibular and/or cerebellar disorders
* Abnormal ophthalmic/optometric disorder (vision disorders)
* Pregnancy
* Serious cardiac disease, malignancy and renal failure

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 participants aged between 18-65 years: 50 female patients who met the ACR 2016 FM diagnostic criteria and 50 pain-free females.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Posture | Baseline
  Posture analysis will be evaluated by DIERS Formetric 4D (Diers International GmbH, Schlangenbad, Germany). Participants will be positioned two meters away from the projector. The slide projector projects a series of parallel light strips on the back of the participant. The back's surface will be captured on camera converted to digital data, and displayed in three dimensions. Every scan will record 12 images over 6 seconds (2Hz) and the manufacturer's recommendations will be followed for processing.
  Spinal reference points, measures of the spinal curves, distance and localization, imbalances of the trunk and pelvis and spinal deviation will be measured. Spine parameters are expressed in millimeters, percentages or degrees depending on the specific parameter.
Balance | Baseline
  The static and dynamic postural control will be measured by HUR SmartBalance BTG4 system (Hur Labs, Tampere, Finland). Participants will be asked to stand barefoot on the balance platform and to stand as quietly as possible, looking forward, during the measurement. While the stable surface is the platform's own floor, the unstable surface is the foam cushion provided by the manufacturer with the device. Data will be collected for 30 seconds. The following parameters will be calculated from the center of pressure (CoP) displacement time series for static postural control: sway area, velocity, Romberg. The limits of stability (LOS) was used to evaluate the dynamic postural control. The participants were asked to tilt their bodies forward, backward, leftward, and rightward for 8 seconds in each direction on the same platform.
Gait | Baseline
  Spatio-temporal gait analysis was performed by Zebris FDM type 3 (Zebris Medical GmbH, Germany) gait analysis system. The system consists of a 3 meters long main platform which contains sensors for measuring the force distributions and a 1 meters long maneuvering platforms that located at the beginning and end of the main platform. Participants will be asked to walk barefoot on the platform. Each participant will walk at their comfortable speed for 2 minutes continuously going from one end to the other along a 5-m walkway in a quiet, well-lit room. The main platform was located in the middle of the system in order to avoid the unstable walking periods on turns. The data were analyzed and recorded on the computer. Foot rotation, stride length, step width, double limb support phase, cadance will be measured. Gait parameters are expressed in centimeters, percentages or degrees depending on the specific parameter.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Baseline
  In FM group; Fibromyalgia Impact Questionnaire (FIQ) will be used to measure the impact of FM on patient's physical function, health status and the severity of disease activity. FIQ is scored from 0-100. Higher scores indicate increased severity of the impact of FM.
Pittsburg Sleep Quality Index (PSQI) | Baseline
  Pittsburg Sleep Quality Index (PSQI) will be used to evaluate sleep quality and the presence of sleep disturbance. The total score consists of 7 components. These components consist of a single question or a combination of several questions. Each question is evaluated on a 0-3 point scale. The total score is between 0-21. A high score indicates poor sleep quality.
Fatigue Severity Scale (FSS) | Baseline
  Fatigue Severity Scale (FSS) will be used to assess fatigue level. The scale consists of 9 questions. Participants are questioned about the level of fatigue in the last week. The questions are scored between 1-7. 1 point: "strongly disagree" and 7 points: "strongly agree", scaled as a Likert-type scale where the degree of agreement increases as the points increase. The highest possible score is 7. Scores of 4 and above indicate pathological fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Baran Tuncer, Medical Doctor, Principal Investigator — Health Sciences University, Ankara Bilkent City Hospital; Selami Akkuş, Prof. Dr., Study Chair — Health Sciences University, Ankara Bilkent City Hospital; İpek Poyraz, Pt., Study Chair — Health Sciences University, Ankara Bilkent City Hospital
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Bilkent/Çankaya, Turkey (Türkiye)

REFERENCES:
- [Result] Sempere-Rubio N, Aguilar-Rodriguez M, Espi-Lopez GV, Cortes-Amador S, Pascual E, Serra-Ano P. Impaired Trunk Posture in Women With Fibromyalgia. Spine (Phila Pa 1976). 2018 Nov 15;43(22):1536-1542. doi: 10.1097/BRS.0000000000002681. PMID 29652782
- [Result] Muto LH, Sauer JF, Yuan SL, Sousa A, Mango PC, Marques AP. Postural control and balance self-efficacy in women with fibromyalgia: are there differences? Eur J Phys Rehabil Med. 2015 Apr;51(2):149-54. Epub 2014 Apr 23. PMID 24755776
- [Result] Heredia Jimenez JM, Aparicio Garcia-Molina VA, Porres Foulquie JM, Delgado Fernandez M, Soto Hermoso VM. Spatial-temporal parameters of gait in women with fibromyalgia. Clin Rheumatol. 2009 May;28(5):595-8. doi: 10.1007/s10067-009-1101-7. Epub 2009 Jan 24. PMID 19169619